CLINICAL TRIAL: NCT00094731
Title: Improving Everyday Memory in At-Risk Elderly
Brief Title: SeniorWISE: Improving Everyday Memory in At-Risk Elderly
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute on Aging (NIA) (NIH)
Allocation: Randomized
Other Study IDs: AG0008; R01AG015384 (NIH)
Record Dates: First submitted 2004-10-21; First posted 2004-10-22 (Estimated); Last update posted 2009-12-11 (Estimated); Status verified 2006-02

CONDITIONS: Aging
Keywords: Aging; Memory; Mental Recall; Mental Processes
MeSH Terms: interventions — Cognitive Training

INTERVENTIONS:
Procedure: Memory Training

SUMMARY:
The purpose of this study is to determine whether classes on memory training will help older adults to improve or maintain their daily activities.

DETAILED DESCRIPTION:
Volunteer participants will be randomly assigned to experimental (memory training) and comparison (health promotion) groups. Both groups will learn strategies for successful aging. Participants will be in the study for 27 months and will be interviewed on five occasions for 3 hours per interview. The classroom-based intervention is an 8-session, 1 1/2 hour course designed to teach older adults the use of strategies to improve everyday memory. Strategically-placed booster sessions will be provided to subjects within 3 months following the last class session.

ELIGIBILITY:
Inclusion Criteria:

* Reside in Austin, Texas or Travis County
* African, Caucasian, or Hispanic heritage
* Fluent in reading and speaking English
* Mini Mental Exam scores of 23-30
* Pass executive function test
* Adequate hearing and vision to enable participation in classroom learning
* Free of Alzheimer's disease or other conditions (e.g., certain cancers) likely to result in mortality before study completion

Exclusion Criteria:

* Under 65
* Score less than 23 on MMSE
* Fail the executive function tests
* Severe sensory losses, hearing or vision, that would prohibit testing or participation
* self-report a diagnosis of Alzheimer's disease or other conditions (e.g., certain cancers) likely to result in mortality before study completion

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 260
Dates: Start 2001-03; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Graham McDougall, PhD, RN, Principal Investigator — University of Texas at Austin, School of Nursing
Locations (1):
- University of Texas at Austin, School of Nursing, Austin, Texas, United States

REFERENCES:
- [Background] McDougall GJ, Montgomery KS, Eddy N, Jackson E, Nelson E, Stark T, Thomsen C. Aging memory self-efficacy: elders share their thoughts and experience. Geriatr Nurs. 2003 May-Jun;24(3):162-8. doi: 10.1067/mgn.2003.43. PMID 12813430
- [Background] McDougall GJ. Memory improvement in octogenarians. Appl Nurs Res. 2002 Feb;15(1):2-10. doi: 10.1053/apnr.2002.29518. PMID 11840404
- [Background] McDougall GJ. I remember that! Building memory confidence in the elderly. Reflect Nurs Leadersh. 2001;27(1):23-5, 45. No abstract available. PMID 11987351
- [Background] Zimmerman T, McDougall GJ Jr, Becker H. Older women's cognitive and affective response to moderate drinking. Int J Geriatr Psychiatry. 2004 Nov;19(11):1095-102. doi: 10.1002/gps.1216. PMID 15481070
- [Background] Austin-Wells V, Zimmerman T, McDougall GJ. ANOPTIMAL DELIVERYFORMATFORPRESENTATIONS TARGETINGOLDER ADULTS. Educ Gerontol. 2003;29(6):493-501. doi: 10.1080/713844396. PMID 18841248
- [Derived] McDougall GJ, Becker H, Acee TW, Vaughan PW, Delville CL. Symptom management of affective and cognitive disturbance with a group of cancer survivors. Arch Psychiatr Nurs. 2011 Feb;25(1):24-35. doi: 10.1016/j.apnu.2010.05.004. Epub 2010 Jul 23. PMID 21251599
- [Derived] McDougall GJ Jr, Becker H, Pituch K, Acee TW, Vaughan PW, Delville CL. The SeniorWISE study: improving everyday memory in older adults. Arch Psychiatr Nurs. 2010 Oct;24(5):291-306. doi: 10.1016/j.apnu.2009.11.001. Epub 2010 Jan 15. PMID 20851321
- [Derived] McDougall GJ Jr, Becker H, Pituch K, Acee TW, Vaughan PW, Delville CL. Differential benefits of memory training for minority older adults in the SeniorWISE study. Gerontologist. 2010 Oct;50(5):632-45. doi: 10.1093/geront/gnq017. Epub 2010 Mar 4. PMID 20203096